CLINICAL TRIAL: NCT04587115
Title: Reducing the Abuse Liability of Prescription Opioids
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Max Eckmann, Associate Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HSC20170141H
Record Dates: First submitted 2020-08-19; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Addiction
Keywords: opioid
MeSH Terms: conditions — Behavior, Addictive | interventions — Risperidone; ziprasidone; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be administered one of two fixed dose drug combinations. The control will be oxycodone plus placebo, whereas the treatment groups will receive oxycodone plus one of the two atypical antipsychotics (Risperidone, Ziprasidone) under study. Study drug will be compounded by outside research pharmacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oxycodone (Placebo Comparator): This arm will be considered the control arm, containing oxycodone as the placebo.
  Interventions: Drug: Oxycodone
- Oxycodone and Risperidone (Experimental): Administration of oxycodone plus risperidone in a single capsule
  Interventions: Drug: Risperidone; Drug: Oxycodone
- Oxycodone and Ziprasidone (Experimental): Administration of oxycodone and risperidone in a single capsule
  Interventions: Drug: Ziprasidone; Drug: Oxycodone

INTERVENTIONS:
Drug: Risperidone — Risperidone 1mg to be used in combination with other drugs
  Other Names: Risperdal
  Arms: Oxycodone and Risperidone
Drug: Ziprasidone — Ziprasidone 80mg to be used in combination with other study drugs
  Other Names: Geodon
  Arms: Oxycodone and Ziprasidone
Drug: Oxycodone — Oxycodone alone in a capsule will be considered the control. Oxycodone 15 mg will also be used in combination with other study drugs
  Other Names: Oxycontin

SUMMARY:
Opioid (commonly called narcotic) pain medicines are, after marijuana, the most commonly abused substances in the United States. Patients who take opioids for legitimate reasons may become addicted; for example, as many as 1 in 4 patients meet the criteria for current opioid dependence. It is very important that a way is found to provide pain relief while minimizing the addiction potential of these widely used pain medications.

The study aim to find out if the use of another type of medication given in addition to an opioid will reduce the addiction potential of the opioid.

The study is trying to find out if the ability of the opioid to relieve pain is changed when given with the other medication, and to see if the euphoric sensation or "liking" of the opioid pain medication is reduced when taken with the other medication.

DETAILED DESCRIPTION:
This study involves the use of an investigational combination of drugs. "Oxycodone with Risperidone" and "Oxycodone with Ziprasidone" are called "Investigational" because the U.S. Food & Drug Administration (FDA) has not approved these drug combinations for the purpose of this study. Individually, each of these drugs is approved by the FDA for other reasons (i.e. oxycodone as a painkiller, while risperidone and ziprasidone are approved as anti-psychotic medications), but the administration of these drugs together has not been studied before or been approved by the FDA for this purpose.

This is the first study involving humans to examine the safety of this combination of drugs and how they work together. The goal of the study is to find out what effects, good and/or bad, it has on people who take them. Because the combination has not been studied in humans before, information about the safety and effectiveness is incomplete and all of the side effects are not yet known.

ELIGIBILITY:
Inclusion Criteria:

* Requirement of prior exposure to opioids

Exclusion Criteria:

* Presence of psychiatric comorbidity
* Presence of chronic pain disorder
* Presence or history of substance use disorder
* Current analgesic or neuroleptic medication usage (any medication for pain, including over-the-counter analgesics like ibuprofen/acetaminophen)
* Pregnancy
* Positive drug urine test
* Continuous opioid misuse measure score of < 9
* Presence or history of diabetes
* Presence or history of cardiac disease or arrhythmia

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of analgesic efficacy- Cold pressor | two weeks
  Perform quantitative evaluations of the analgesic efficacy of a novel fixed dose combination (FDC) of an opioid (oxycodone) in combination with one of two atypical antipsychotic drugs (either risperidone or ziprasidone) compared to the opioid alone. Analgesic efficacy will be measured with the cold pressor task which measures thermal pain. The cold pressor task measures the time the participant can tolerate their hand being submerged in the cold water up to a maximum of 5 minutes.

SECONDARY OUTCOMES:
Evaluation of analgesic efficacy- Thumb pressor | two weeks
  Perform quantitative evaluations of the analgesic efficacy of a novel fixed dose combination (FDC) of an opioid (oxycodone) in combination with one of two atypical antipsychotic drugs (either risperidone or ziprasidone) compared to the opioid alone. Analgesic efficacy will be measured with the thumb pressor task which measures mechanical pain. The thumb pressor task measures the amount of weight they can tolerate on the nail of their thumb up to a maximum of 10 kg.
Drug liking | two weeks
  Examine subjective ratings of drug liking of the FDC compared to that of the opioid alone using the Bipolar Visual analog scale on a scale of 0-Dislike to 100-Extremely like.
Addiction Research Center Inventory test questionnaire | two weeks
  Perform the Addiction Research Center Inventory Short Form (ARCI-SF) questionnaire to assess the drug-induced transient alterations in distinct mood states of the FDC compared to those of the opioid alone. The ARCI is a self-administered, standardized questionnaire for assessing subjective effects of psychoactive drugs that was developed in the early 1960s at the National Institute of Mental Health Addiction Research Center. For this study, the study team will be using the 49-item short form. Outcome will be assessed using categorical and continuous data analysis comparing across groups. The ARCI-SF measures the subjective effects of a variety of drugs such as alcohol, morphine, LSD, and pentobarbital by a score for each subset. The higher a participant scores on a subset, the more similar the effects of the drug are to the known drug such as alcohol.
Profile of Mood States test questionnaire | two weeks
  Perform a subset of the Profile of Mood States questionnaire to assess drug-induced transient alterations in distinct mood states following administration of the FDC compared to those of the opioid alone. POMS is a self-administered, standard validated psychological test formulated by McNair et al. (1971). It is a used to assess transient, distinct mood states. The questionnaire contains 65 words/statements that describe feelings people have. Outcome will be assessed using categorical and continuous data analysis comparing across groups. The POMS is a non-diagnostic test that assesses transient and distinct mood states such as tension, depression, anger, fatigue, confusion, vigor, and total mood disturbance. The higher a participant scores in each group, the more they experience that mood state.

CONTACTS AND LOCATIONS:
Overall Officials: Max Eckmann, MD, Principal Investigator — University of Texas Health at San Antonio
Locations (1):
- Westgate Pain Clinic, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared with other collaborating investigators, and unidentified data will be shared at study completion as a publication.
Supporting Information: Study Protocol, SAP
Time Frame: At study completion.